CLINICAL TRIAL: NCT01540604
Title: An Open-label, Un-controlled, Single-centre Trial Investigating the Efficacy and Safety of CRD007 in Children With Duchenne Muscular Dystrophy (DMD) or Becker Muscular Dystrophy (BMD) or Children Being Symptomatic Carriers for DMD or BMD
Brief Title: CRD007 for the Treatment of Duchenne Muscular Dystrophy, Becker Muscular Dystrophy and Symptomatic Carriers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RSPR Pharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Cardoz-004
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
Keywords: DMD; BMD; symptomatic carriers
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

ARMS (1):
- CRD007 10 mg tablet (Experimental)
  Interventions: Drug: CRD007

INTERVENTIONS:
Drug: CRD007

SUMMARY:
This is an investigation of the efficacy and safety of CRD007 in Duchenne Muscular Dystrophy (DMD), Becker Muscular Dystrophy (BMD) and symptomatic carriers.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dystrophinopathy

Exclusion Criteria:

* Severe functional impairment

Ages: 2 Years to 11 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: T Sejersen, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Stockholm, Sweden